CLINICAL TRIAL: NCT06852924
Title: A Single-center Prospective Randomized Controlled Trial of Inhaled Nitric Oxide in the Treatment of High Amplitude Pulmonary Edema(HAPE)
Brief Title: Inhaled Nitric Oxide for High Amplitude Pulmonary Edema (HAPE)
Acronym: HAPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Novlead Inc. (Industry)
Collaborators: Tibet Fokind Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAPE23-06
Record Dates: First submitted 2025-02-14; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: High Altitude Pulmonary Hypertension
Keywords: iNO; HAPE
MeSH Terms: conditions — Pulmonary edema of mountaineers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group: Received traditional treatment (No Intervention): Control group: received traditional treatment, intravenous injection of furosemide, aminophylline, dexamethasone, oxygen inhalation, and other symptomatic treatment drugs.
- Inhaled Nitric Oxide (iNO) - Group A (Experimental): On the basis of traditional treatment, NO 15 ppm was inhaled 30min/ time, twice/day, once in the morning and once in the afternoon.
  Interventions: Device: Nitric Oxide Generation and Delivery System
- Inhaled Nitric Oxide (iNO)-Group B (Experimental): On the basis of traditional treatment, NO 15 ppm was inhaled 2h/ time, twice/day, once in the morning and once in the afternoon.
  Interventions: Device: Nitric Oxide Generation and Delivery System

INTERVENTIONS:
Device: Nitric Oxide Generation and Delivery System — The Nitric Oxide Generation and Delivery System is used to deliver nitric oxide for inhalation therapy into the inspiratory limb of the patient breathing circuit in a way that provides a constant concentration of nitric oxide (NO), as set by the user, to the patient throughout the inspired breath.
  Arms: Inhaled Nitric Oxide (iNO) - Group A; Inhaled Nitric Oxide (iNO)-Group B

SUMMARY:
High Altitude Pulmonary Edema (HAPE) is a critical, non-cardiogenic pulmonary edema that manifests in high-altitude conditions, marked by the rapid onset of symptoms such as dyspnea, cough, frothy sputum, and cyanosis. It represents a significant cause of mortality among high-altitude illnesses due to its swift progression and elevated fatality rates if not addressed promptly. The pathophysiological mechanisms underlying HAPE include excessive hypoxic pulmonary vasoconstriction, increased permeability of the pulmonary vasculature, impaired clearance of fluid from the lungs, and systemic fluid retention. A pivotal factor in HAPE is pulmonary arterial hypertension (PAH), characterized by a progressive rise in pulmonary arterial pressure and resistance, which can ultimately lead to right heart failure. Recent developments in the management of HAPE have introduced inhaled nitric oxide (iNO) as a selective pulmonary vasodilator, which effectively lowers pulmonary arterial pressure and enhances oxygenation without inducing systemic hypotension. The INOwill N300 device, created by Nanjing Novlead Biotech, is a portable iNO delivery system that produces nitric oxide gas on-site, thereby obviating the need for gas cylinders. This device also facilitates real-time monitoring of nitric oxide, nitrogen dioxide, and oxygen concentrations, ensuring safe and effective treatment. This innovative strategy shows potential for improving clinical outcomes in patients with HAPE while addressing logistical challenges encountered in high-altitude environments.

DETAILED DESCRIPTION:
This study utilized the inaugural nitric oxide therapeutic device sanctioned by the State Drug Administration, which possesses independent intellectual property rights (INOwill N300, Nanjing Novlead Biotechnology Co., LTD.). The device is compact and generates nitric oxide gas upon activation, eliminating the need for cylinders for the storage and transport of nitric oxide. It employs an electrochemical catalytic reduction method to produce nitric oxide gas in real-time and automatically administers the gas to the respiratory circuit at a predetermined concentration, based on flow monitoring. The phase change sensor sampling technology enables real-time monitoring of the concentrations of nitric oxide, nitrogen dioxide, and oxygen at the patient end of the respiratory circuit, thereby ensuring the safety of clinical interventions.

The primary aim of this investigation was to assess the efficacy of inhaled nitric oxide (iNO) in the management of mild to moderate high altitude pulmonary edema (HAPE) in comparison to a control group. Key parameters evaluated included the onset time of changes in oxygenation, the duration until symptom resolution (as measured by the Lake Louise Acute Mountain Sickness score), the time required for improvement in imaging indicators, and the proportions of patients categorized as cured, effective, ineffective, or experiencing severe HAPE by days 3 to 7 of treatment. Additionally, the length of hospital admission or stay was recorded for patients receiving iNO therapy for high altitude pulmonary edema. This study aimed to elucidate the impact of iNO on enhancing oxygenation and pulmonary circulation in patients with high altitude pulmonary edema relative to the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged between 18 and 65 years.
2. A score on the Lake Louise Acute Mountain Sickness Scale ranging from 3 to 9 points, as outlined in Annex 2, recorded in 2018.
3. Chest X-ray findings that demonstrate either thickening of the lung texture bilaterally or the presence of nodular opacities in the lower regions of both lungs.
4. Capacity to provide informed consent in accordance with local regulatory requirements.

Exclusion Criteria:

1. Confirmed contraindications for the use of nitric oxide include the following (refer to "5.3.4 NO Contraindications"):

   * Severe hypoplasia of the left heart or duct-dependent congenital heart disease;
   * Life-threatening congenital anomalies and congestive heart failure;
   * Congenital methemoglobinemia;
   * Severe hemorrhagic conditions, including intracranial hemorrhage, intraventricular hemorrhage, and pulmonary hemorrhage.
2. Severe left ventricular dysfunction, characterized by a left ventricular ejection fraction (LVEF) of less than 40%.
3. Pulmonary edema resulting from other cardiac, pulmonary, thoracic, or systemic disorders.
4. Coexistence with high altitude cerebral edema.
5. A history of lung malignancy, lung resection, or lung transplantation.
6. Barotrauma, which may include pneumothorax, subcutaneous and mediastinal emphysema, or the presence of a closed drainage tube in the thoracic cavity.
7. Clinically significant or persistent thrombocytopenia, defined as a platelet count of less than 50×10^9/L.
8. Administration of pulmonary hypertension medications, such as sildenafil, bosentan, or prostacyclins, within the preceding 30 days.
9. Noncompliance with study protocols and unwillingness to provide informed consent.
10. Any other conditions that the clinician deems render the subject unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Oxygen Index | Through study completion, an average of 5 days
  The change of oxygenation index (PaO2 or SpO2/FiO2) from baseline, and the time required for oxygenation index to improve by ≥20%

SECONDARY OUTCOMES:
Progression of HAPE | Through study completion, an average of 5 days
  The proportion and time of HAPE cured, markedly effective, ineffective, or severe
Symptoms Improvement | Through study completion, an average of 5 days
  Change of symptom improvement (Lake Louise AMS score, vital signs, imagings)
Hospital Stays | Through study completion, an average of 5 days
  The length of hospital stay compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Jingxin Cao, Principal Investigator — Tibet Fokind Hospital
Locations (1):
- Tibet Fokang Hospital, Lhasa, Tibet, China